CLINICAL TRIAL: NCT05792397
Title: A Multicenter Prospective Single-arm Study to Evaluate the Safety and Efficacy of a Novel Transcatheter Pulmonary Thrombectomy System Which Named 'TwiFlow' for Acute Pulmonary Embolism
Brief Title: TwiFlow Thrombectomy Catheter sYstem for Acute Pulmonary Embolism (Twi-TYPE Study)
Acronym: Twi-TYPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Morningside (Nantong) Medical Co.,Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHENXING-2022-05
Record Dates: First submitted 2023-03-05; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Acute Pulmonary Embolism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): The arm contains patients with acute pulmonary embolism who undergoing interventional therapy with transcatheter pulmonary embolectomy system which named 'TwiFlow-Thrombectomy Catheter System'
  Interventions: Device: TwiFlow-Thrombectomy Catheter System

INTERVENTIONS:
Device: TwiFlow-Thrombectomy Catheter System — Patients with acute pulmonary embolism and meeting the conditions of this clinical trial will accept the pulmonary embolism removal operation by the novel device named 'TwiFlow-Thrombectomy Catheter System'

SUMMARY:
As a multicenter prospective single-arm clinical study, the investigators plan to recruit patients with acute pulmonary intravascular embolization from nationwide multi-center hospital organizations in China. The investigators use the production of transcatheter pulmonary artery bolt system which named 'TwiFlow Thrombectomy Catheter System' developed by the MorningSide (NanTong) medical device Co., LTD. on pulmonary artery interventional therapy to evaluating the efficacy and safety of this novel system in the treatment of patients with pulmonary intravascular embolization disease.

DETAILED DESCRIPTION:
As a multicenter prospective single-arm clinical study, the investigators plan to evaluate the new production's efficacy and safety which named 'TwiFlow-Thrombectomy Catheter System'. This study will be carried out in nationwide multi-center hospital organizations in China. According to the statistical principle, the sample size of this study was estimated, and the final number of selected cases was 127. After screening, all subjects will be treated with transcatheter pulmonary artery thrombectomy system, and clinical follow-up will be conducted at 48 hours, 14 days and 30 days after surgery. Right Ventricular/Left Ventricular decline from baseline to 48 hours after surgery and the incidence of major adverse events (MAE) within 48 hours after surgery were used as primary endpoints. In instrument performance evaluation, the success rate of surgery, postoperative immediate target lesion embolus removal efficiency, pulmonary artery pressure changes before and after operation value, values of arterial oxygen partial pressure changes before and 14 days after operation, death rates related to the equipment in 48 hours after surgery, incident rate of bleeding in 48 hours after operation, postoperative clinical deterioration rate in 48 hours after surgery, postoperative pulmonary vascular injury incidence in 48 hours after surgery, the incidence of heart damage injury in 48 hours after surgery, all-cause death rate in 30 days after surgery, and symptomatic Pulmonary Embolization recurrence rate in 30 days after surgery were secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. 18≤ age ≤75, no gender limitation;
2. patients clinically diagnosed as acute pulmonary embolism requiring pulmonary artery thrombosis clearance;
3. RV/LV ratio ≥0.9;
4. Duration of pulmonary embolism symptoms ≤14 days
5. Systolic blood pressure ≥90mmHg
6. Patients who agreed to participate in the study and voluntarily signed the informed consent.

Exclusion Criteria:

1. Target vessel diameter < 6.6mm;
2. Calcification, plaque or stenosis of target lesions;
3. Pulmonary arterial hypertension with peak pulmonary arterial pressure >70mmHg;
4. Vasopressor is required after infusion to maintain pressure ≥90mmHg;
5. Hematocrit < 28%;
6. Patients with left bundle branch block;
7. A history of chronic left heart failure and left ventricular ejection fraction≤30%;
8. Patients with abnormal renal function (serum creatinine > 1.8 mg/dL or >159umol/L);
9. Patients with known coagulopathy or bleeding tendency (platelet<100×109/L, or INR> 3);
10. Patients who cannot receive antiplatelet or anticoagulant therapy;
11. Patients who underwent cardiovascular or pulmonary open surgery within 7 days before surgery;
12. Patients with intracardiac thrombosis;
13. Patients treated with extracorporeal membrane oxygenation;
14. Patients known to be allergic to contrast agents;
15. Patients with diseases that may cause difficulty in treatment and evaluation (such as malignant tumor, acute infectious disease, sepsis, general condition that cannot tolerate surgery, life expectancy less than 3 months, etc.);
16. Pregnant and lactating women;
17. Patients who are participating in clinical trials of other drugs or medical devices;
18. Other patients deemed unsuitable for the study by the investigator;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Right Ventricular/Left Ventricular decline from baseline to 48 hours after surgery | before and 48 hours after surgery
  Right Ventricular (RV) and Left Ventricular (LV) were recorded during the screening period and 48 hours after surgery by echocardiography or pulmonary artery CT (CTPA), and RV/LV and RV/LV reduction were calculated. The target RV/ LV reduction from baseline to 48 hours after surgery was at least 0.2.
The incidence of major adverse events (MAE) within 48 hours after surgery | 48 hours after surgery
  The incidence of major adverse events (MAE) during and 48 hours after surgery was observed and recorded, and the incidence of MAE was calculated (referring to the definition of MAE). The target incidence of MAE 48 hours after surgery was less than 25%.
  MAE events defined as those occurring within 48 hours of treatment include device-related death, massive bleeding, pulmonary vascular injury, and cardiac injury.
  Haemorrhage: Disabling or life-threatening bleeding, or severe haemodynamic injury.
  Pulmonary vascular injury: Defined as perforation or injury of a major pulmonary artery branch requiring surgical open surgical intervention.
  Cardiac injury: Defined as heart injury requiring surgical open surgical intervention.

SECONDARY OUTCOMES:
instrument performance evaluation | intraoperative period
  researchers try to evaluate the twi-system instrument' performance during the operation, so investigators will review whether the device system successfully performed the following steps: 1.Pulmonary thrombectomy system transport to the thromboembolic site (yes or not), 2.The thrombectomy stent was successfully deployed (yes or not), 3.the clot-plug is retracted successfully (yes or not), 4. the thrombectomy device safely removed from the body (yes or not), 5. Thrombus suction catheter delivers to the specified thromboembolic location (yes or not), 6.the thrombus suction catheter delivery system safely removed from the body (yes or not). The study predefine the answer"yes" to 1 point and "no" to 0 point, then investigators will calculate the total scores according above 6 steps and evaluate the twi-system instrument' performance during the operation.
the success rate of surgery | intraoperative period
  Surgical success was defined as successful thrombectomy without MAE.
pulmonary artery pressure changes before and after operation value | before the pulmonary intravascular embolization removal procedure began and after the embolization removal operation end immediately
  Changes in pulmonary artery pressure before and after operation = postoperative pulmonary artery pressure - preoperative pulmonary artery pressure
values of arterial oxygen partial pressure changes before and after operation | before the pulmonary intravascular embolization removal procedure began and 14 days after surgery
  Preoperative and postoperative arterial oxygen partial pressure = 14 days postoperative arterial oxygen partial pressure - preoperative arterial oxygen partial pressure
postoperative clinical deterioration rate in 48 hours after surgery | 48 hours after surgery]
  Clinical deterioration include instrumentation related events such as unplanned endotracheal intubation, mechanical ventilation, arterial hypotension (>1 hour) or shock, cardiopulmonary resuscitation, significant deterioration of oxygenation, and emergency surgical embolectomy.
all-cause death rate in 30 days after surgery | 30 days after surgery
  all-cause death
symptomatic Pulmonary Embolization recurrence rate in 30 days after surgery | 30 days after surgery
  patients occur pulmonary embolism again and represent related clinical symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Zhuang Hui, Dr., Study Chair — Xiamen Cardiovascular Hospital, Xiamen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moore K, Kunin J, Alnijoumi M, Nagpal P, Bhat AP. Current Endovascular Treatment Options in Acute Pulmonary Embolism. J Clin Imaging Sci. 2021 Jan 25;11:5. doi: 10.25259/JCIS_229_2020. eCollection 2021. PMID 33598362
- [Result] Villalba L, Nguyen T, Feitosa RL Jr, Gunanayagam P, Anning N, Dwight K. Single-session catheter-directed lysis using adjunctive power-pulse spray with AngioJet for the treatment of acute massive and submassive pulmonary embolism. J Vasc Surg. 2019 Dec;70(6):1920-1926. doi: 10.1016/j.jvs.2019.03.038. Epub 2019 May 27. PMID 31147112
- [Result] Al-Hakim R, Bhatt A, Benenati JF. Continuous Aspiration Mechanical Thrombectomy for the Management of Submassive Pulmonary Embolism: A Single-Center Experience. J Vasc Interv Radiol. 2017 Oct;28(10):1348-1352. doi: 10.1016/j.jvir.2017.06.025. PMID 28941516
- [Result] Sista AK, Horowitz JM, Tapson VF, Rosenberg M, Elder MD, Schiro BJ, Dohad S, Amoroso NE, Dexter DJ, Loh CT, Leung DA, Bieneman BK, Perkowski PE, Chuang ML, Benenati JF; EXTRACT-PE Investigators. Indigo Aspiration System for Treatment of Pulmonary Embolism: Results of the EXTRACT-PE Trial. JACC Cardiovasc Interv. 2021 Feb 8;14(3):319-329. doi: 10.1016/j.jcin.2020.09.053. Epub 2021 Jan 13. PMID 33454291
- [Result] Wible BC, Buckley JR, Cho KH, Bunte MC, Saucier NA, Borsa JJ. Safety and Efficacy of Acute Pulmonary Embolism Treated via Large-Bore Aspiration Mechanical Thrombectomy Using the Inari FlowTriever Device. J Vasc Interv Radiol. 2019 Sep;30(9):1370-1375. doi: 10.1016/j.jvir.2019.05.024. Epub 2019 Jul 30. PMID 31375449
- [Result] Yasin JT, Davis R, Saemi A, Regunath H, Krvavac A, Saboo SS, Bhat AP. Technical efficiency, short-term clinical results and safety of a large-bore aspiration catheter in acute pulmonary embolism - A retrospective case study. Lung India. 2020 Nov-Dec;37(6):485-490. doi: 10.4103/lungindia.lungindia_115_20. PMID 33154209
- [Result] Tu T, Toma C, Tapson VF, Adams C, Jaber WA, Silver M, Khandhar S, Amin R, Weinberg M, Engelhardt T, Hunter M, Holmes D, Hoots G, Hamdalla H, Maholic RL, Lilly SM, Ouriel K, Rosenfield K; FLARE Investigators. A Prospective, Single-Arm, Multicenter Trial of Catheter-Directed Mechanical Thrombectomy for Intermediate-Risk Acute Pulmonary Embolism: The FLARE Study. JACC Cardiovasc Interv. 2019 May 13;12(9):859-869. doi: 10.1016/j.jcin.2018.12.022. PMID 31072507